CLINICAL TRIAL: NCT06155578
Title: Randomized Placebo-controlled Trial of the Safety and Efficacy of Topical Sodium Metabisulfite for the Treatment of Calcinosis in Patients With Systemic Sclerosis.
Brief Title: Safety and Efficacy of Topical Sodium Metabisulfite for the Treatment of Calcinosis in Patients With Systemic Sclerosis
Acronym: Cal-23
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Liga Panamericana de Asociaciones de Reumatologia (PANLAR) (Other)
Responsible Party: Principal Investigator, Antonia Valenzuela, MD, MS, Assistant Professor at Pontificia Universidad Católica de Chile, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 220421002
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Systemic Sclerosis; Calcinosis
Keywords: Systemic Sclerosis; calcinosis; sodium metabisulfite; topical
MeSH Terms: conditions — Scleroderma, Systemic; Calcinosis | interventions — sodium metabisulfite

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial with subjects allocated to topical 25% sodium metabisulfite or placebo cream twice daily.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research products will be prepared in pediatric cold cream (water in oil emulsion) at a concentration of 25% or placebo, with identical packing and labeling, each identified by an exclusive number ID which will be assigned by a researcher not involved with the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium metabisulfite cream (Active Comparator): Sodium metabisulfite prepared in pediatric cold cream (water in oil emulsion) at a concentration of 25% to be applied on calcinosis topically twice daily.
  Interventions: Drug: Topical 25% sodium metabisulfite (SM) in pediatric cold cream
- Placebo cream (Placebo Comparator): Pediatric cold cream (water in oil emulsion) to be applied on calcinosis topically twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical 25% sodium metabisulfite (SM) in pediatric cold cream — Topical 25% sodium metabisulfite (SM) in pediatric cold cream will be applied twice daily on hand calcinosis.
  Other Names: cold cream
  Arms: Sodium metabisulfite cream
Drug: Placebo — Pediatric cold cream will be applied twice daily on hand calcinosis.
  Other Names: cold cream
  Arms: Placebo cream

SUMMARY:
This prospective placebo-controlled trial will enroll 20 patients with SSc and at least one calcinotic lesion of the hands that is palpable on physical examination and measurable on hand radiographs. Each subject will undergo a screening evaluation 1 month before treatment with the study drug is initiated. Each subject will be instructed to blindly self-apply either topical 25% sodium metabisulfite or placebo cream twice daily. In-person follow-up evaluations will be performed after 4-months, with monthly telehealth follow-up visits to ensure adherence and arrange study drug refill deliveries.

DETAILED DESCRIPTION:
1. Background:

   Calcinosis cutis is the deposition of calcium in the skin and subcutaneous tissues. It is a common and debilitating manifestation of systemic sclerosis (SSc), affecting 1 in 4 of these patients over the course of their disease. Calcinosis in SSc occurs most frequently in the hands, particularly the fingers, and within the fingers, most commonly in the thumbs or index of the dominant hand. Calcinosis in SSc can cause pain, soft tissue swelling around the calcium deposits, ulcers with superimposed infection, or deformities, leading to significant impact on quality of life.

   Treatment for calcinosis cutis is often difficult and unsuccessful and remains an unmet need in patients with SSc. Evidence mainly comes from small retrospective studies, case series, and case reports, since no large, prospective randomized controlled trials have been conducted. The response to various agents, such as topical or oral aluminum hydroxide, topical or intralesional sodium thiosulfate, intralesional corticosteroids, calcium-channel blockers, minocycline, bisphosphonates, and surgical excision has remained largely unsatisfactory.

   Topical, intralesional and intravenous (IV) sodium thiosulfate have been studied as treatments for disorders of cutaneous calcium deposition. The mechanism of sodium thiosulfate in the treatment of calcium-related disorders is thought to be multifactorial. It is believed to act by transforming calcium into calcium thiosulfate salts, thus increasing calcium solubility. In addition, it may increase the production of hydrogen sulfide, which has vasodilatory, antioxidant and anti-inflammatory properties, and may cause direct inhibition of vascular calcifications.

   Sodium metabisulfite (SM) is an inorganic compound used as a disinfectant, antioxidant and preserving agent that, when reacting with oxygen, becomes sodium sulfate, a metabolite of sodium thiosulfate that has a similar ability to inhibit calcium oxalate agglomeration and calcium stone formation. In 2016, topical 25% SM was used for the first time in four patients with dystrophic calcinosis cutis (one with SSc, two with dermatomyositis and one with radio-dermatitis after breast cancer), showing signiﬁcant decrease in size, erythema, and pain. The authors hypothesized that topical SM may dissolve calcium deposits and promote local vasodilation and wound healing. Since then, topical sodium metabisulﬁte use has been reported as an inexpensive, safe and promising new agent for the treatment of calcinosis cutis.

   On behalf of the Scleroderma Clinical Trial Consortium (SCTC) Calcinosis Working Group, we developed and validated a novel radiographic scoring system to assess the severity of calcinosis affecting the hands of patients with SSc that accounts for area coverage, density, and anatomic location. This scoring system is feasible and was found to have excellent intra- and inter-rater reliability with intra-class correlation coefficients (ICC) of .93 (.89-.97) and .89 (.86-.92), respectively. We confirmed the excellent inter-rater reliability of our radiographic calcinosis scoring system and demonstrated its usefulness to detect change over time in a recent study of 39 patients and a validation cohort of 19 patients.Calcinosis in SSc usually progresses over time. In this same study, 80% of patients had worsening or unchanged calcinosis without treatment at 1 year follow-up as measured by this radiologic scoring system.

   Given that calcinosis is a frequent, debilitating, and progressive complication of SSc with no effective therapies, a clinical trial, using novel outcome measures, testing the safety and efficacy of a potential treatment of calcinosis is warranted.
2. Primary/Secondary objectives:

   Our main objective is to conduct a study with the following primary and secondary endpoints.

   Primary endpoints:
   * To assess the safety and tolerability of using topical 25% SM applied twice daily in SSc patients with calcinosis affecting the hands.
   * To assess the efficacy of topical 25% SM versus placebo in stabilizing the calcinosis burden or reducing the radiographic progression of calcinosis over four months.

   Secondary endpoints:
   * To assess the effect of topical 25% SM on the change in the Mawdsley Calcinosis Questionnaire, and patient and physician assessment of calcinosis severity over four months.
   * To assess the effect of topical 25% SM on the change in size of calcinosis on ultrasound.

   To assess the presence of markers of vascular damage by tape stripping in SSc patients with calcinosis.
3. Hypothesis:

   We hypothesize that topical SM may be beneficial in the treatment of calcinosis in patients with SSc stabilizing the burden of calcinosis as measured by the SCTC radiologic scoring system.
4. Study design:

   This prospective placebo-controlled trial will enroll 20 patients with SSc and at least one calcinotic lesion of the hands that is palpable on physical examination and measurable on hand radiographs. Each subject will undergo a screening evaluation 1 month before treatment with the study drug is initiated. Each subject will be instructed to blindly self-apply either topical 25% SM or placebo cream twice daily. Follow-up in-person evaluations will be performed a 4-month period, with monthly telehealth follow-up visits to ensure adherence and provide study drug.
5. Study population:

   The population for this study will consist of adult SSc patients with evidence of at least one calcinotic lesion of the hands that is palpable on physical examination and measurable on hand radiographs. Inclusion and exclusion criteria have been entered elsewhere.
6. Description of the treatment:

   Each subject will be randomized and instructed to blindly self-apply, either SM prepared in pediatric cold cream (water in oil emulsion) at a concentration of 25% or placebo topically twice daily, which will be continued as tolerated. Vinyl gloves will be supplied to each patient to improve topical absorption. Patients will participate in a learning session with examples and instructions on how to use the cream. Detailed instructions will be provided to patients for their reference during treatment.
7. Description of Assessments:

   Medical history including SSc: Significant past or present illnesses, current prescription, or nonprescription medications (including vitamins and herbal products), and history of allergies or idiosyncratic responses to drugs will be noted at the time of enrolment. Demographic and clinical data, including age, gender, race, smoking status, disease duration defined from onset of RP and from first non-RP symptom, SSc skin subtype, internal organ involvement, and auto-antibodies including SSc-specific and anti-phospholipid antibodies will be recorded.

   Physical examination: A complete physical examination will be conducted by a physician at screening, baseline and at end of study.

   Vital Signs: Systolic and diastolic blood pressure, heart rate, and temperature (°C) will be measured after sitting for 5 minutes at screening, baseline, and 4 months. Vital signs should also be assessed in the case of abnormal clinical signs and symptoms.

   Laboratory tests: Blood and urine samples for the measurement and evaluation of routine blood laboratory test CBC, CMP, and pregnancy urine test for fertile women will be collected at screening and at the end of the study.

   Tape stripping: Skin samples will be obtained using the tape stripping technique, utilizing five standard D-Squame® sampling discs (Cuderm, Dallas, USA) at the same site on the hands before the initiation of topical treatment with SM or a placebo and at the conclusion.

   Radiological examination of calcinosis: Descripcion has been entered elsewhere

   Ultrasonography (US): Descripcion has been entered elsewhere.

   Mawdsley Calcinosis Questionnaire (MCQ): Descripcion has been entered elsewhere.

   Patient and Physician global assessments: Descripcion has been entered elsewhere.
8. Safety monitoring and reporting Safety: During the study, the primary assessment of safety will be the development of adverse events.

   Adverse Event (AE): An AE is any untoward medical experience occurring to a subject during a clinical trial whether it is related to the study drug. An AE may include an intercurrent illness, injury, or any other concomitant impairment of the subject's health, as well as abnormal laboratory findings if deemed to have clinical significance. AEs may also include worsening of an existing symptom or condition or post-treatment events that occur because of protocol-mandated procedures.

   Severe Adverse Event (SAE): A SAE is an AE occurring at any dose that results in any of the following outcomes:
   * Death
   * A life-threatening AE
   * Inpatient hospitalization or prolongation of existing hospitalization
   * A persistent or significant disability / incapacity
   * A congenital anomaly / birth defect

   In addition, important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the subject and require medical / surgical intervention to prevent one of the outcomes listed above.
9. Statistical Considerations:

   Statistical analysis:

   Descriptive statistics and frequency distributions of all variables of interest will be reported as proportions (%) for categorical variables and as mean ± standard deviation or median (range) for continuous variables. Baseline to 4-month differences and 95% confidence intervals will be calculated for scored outcomes (x-ray score, physician's global assessment by VAS, and quality of life measurements). For the primary efficacy endpoint, mean change and standard deviation in calcinosis burden assessed by radiograph from baseline to 4-month visit, we will use Student's t-test. The mean rate of change of calcinosis in radiograph will be calculated with the following formula: (Year 1 XR score - Baseline XR score)/time. XR score is defined as: sum of scores for 22 weighted areas affecting each hand: %area coverage (0-100) X density (1-3) X weight for each area.(19)

   Sample size calculation:

   We are planning a study of a continuous response variable from independent control and experimental subjects with 1 control(s) per experimental subject. In a previous study the response within each subject group was normally distributed with standard deviation 3,2. If the true difference in the experimental and control means is 4,2, we will need to study 10 experimental subjects and 10 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0,8. The Type I error probability associated with this test of this null hypothesis is 0,05.
10. Risks of Treatment The main risks of the treatment are the same as those secondary to the use of any other cream or topical treatment; participants may experience burning, pain, or allergies in the treatment area. In case of any of these adverse effects, the participant will be evaluated by a Dermatologist member of our team.

However, in a 2022 review in which the best scientific evidence of all published works that included the use of sodium metabisulfite cream for the treatment of skin calcifications in autoimmune patients was analyzed, out of a total of 7 patients, none of them presented any adverse effect with the application of said cream, so with the current evidence to date, the probability of presenting any adverse effect from the use of this topical treatment is very low, that is, less than 0.1% or less than 1 person in every 1000 people who use this cream.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age > 18 years of age
* Diagnosis of limited or diffuse cutaneous systemic sclerosis (SSc) according to the revised 2013 ACR/EULAR classification criteria for SSc (21)
* Radiological and physical examination evidence of at least one subcutaneous calcium deposition in the hands that is clinically apparent as part of routine clinical care.
* If female of childbearing potential, the patient must have a negative pregnancy test at screening and baseline visits
* Oral corticosteroids (≤ 5 mg/day of prednisone or equivalent) and NSAIDs are permitted if the patient is on a stable dose regimen for ≥ 2 weeks prior to screening and throughout the study
* Oral CCB, alpha-1-antagonists, ACE-inhibitors, angiotensin receptor blockers, and protein-pump inhibitors are permitted if the doses are stable for 4 weeks prior to screening and throughout the study.

Exclusion Criteria:

* Rheumatic disease other than SSc
* Allergy to sodium metabisulfite
* Pregnant or nursing women
* Concurrent malignancy except non-melanoma skin cancers
* Patients receiving bisphosphonates, warfarin, colchicine, minocycline, intravenous immunoglobulins, or biological agents specifically abatacept or rituximab within 4 weeks of screening
* Patients receiving local treatments for calcinosis of the hands including surgical removal or intralesional steroid injections within 12 weeks of screening or throughout the study.
* Patients who have participated in another clinical trial of an investigative agent within 30 days of screening (or 5 half-lives of the investigational drug, whichever is longer)
* Patients with a history of drug or alcohol abuse within 6 months of screening
* Any medical condition that, in the opinion of the investigator, might interfere with the subject's participation in the study or poses an added risk for the subject
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of using topical 25% SM applied twice daily in SSc patients with calcinosis affecting the hands | 4 months
  The primary assessment of safety will be the development of adverse events. Any significant changes to the subject's medical condition, physical examination, and concomitant medications will be documented throughout the course of the study. Any untoward medical experience will be recorded as an adverse event.
To assess the efficacy of topical 25% SM versus placebo in stabilizing the calcinosis burden or reducing the radiographic progression of calcinosis over four months. | 4 months
  Radiograph of the hands will be scored using the SCTC radiographic calcinosis scroing system

SECONDARY OUTCOMES:
To assess the effect of topical 25% SM on the change in the Mawdsley Calcinosis Questionnaire, and patient and physician assessment of calcinosis severity over four months. | 4 months
  The MCQ is a novel patient reported outcome measure developed to assess the severity and impact of SSc-related calcinosis in clinical studies/clinical practice. The content of this questionnaire is patient-generated and includes 17 questions related to the impact of calcinosis rated from 0 (no limitation) to 10 (worst limitation possible), organized in 6 items of quantification of calcinosis, a test question of interpretation and 3 domains: Pain/sensation (5 items); Physical Function (4 items) and Psychological Impact (6 items). Patients will fill up the MCQ at baseline and 4 months.
To assess the effect of topical 25% SM on the change in size of calcinosis on ultrasound. | 4 months
  US is a rapid and noninvasive technique that can provide in-vivo information for the detection and monitoring of calcium depositions. (25) Calcinosis in US can be identified as hyperechoic lesions with or without shadowing, located in the skin, soft tissue, tendons, peritendinous or periarticular areas. Length, width, and depth of calcinotic deposits will be measured in millimeters (mm) at baseline and 4 months using high-frequency color Doppler ultrasound examination.
To assess the presence of markers of vascular damage and inflammation by tape stripping in SSc patients with calcinosis. | 4 months
  Tape stripping is a non-invasive and largely used technique. The sampling of consecutive subcutaneous layers by means of glues on tapes allows to evaluate the composition of the skin, and to study the development of inflammatory mediators, wound healing, and other processes.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Valenzuela, MD, MS, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Antonia Valenzuela, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Will be considered upon reasonable request.
Supporting Information: Study Protocol
Time Frame: End of study
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Ricardo JW, Sun HY, Gorji M, Sebaratnam DF. Topical sodium thiosulfate as treatment of calcinosis cutis: Case series and systematic review. J Am Acad Dermatol. 2022 Aug;87(2):443-444. doi: 10.1016/j.jaad.2021.09.013. Epub 2021 Sep 16. No abstract available. PMID 34537249
- [Background] Valenzuela A, Baron M; Canadian Scleroderma Research Group; Herrick AL, Proudman S, Stevens W; Australian Scleroderma Interest Group; Rodriguez-Reyna TS, Vacca A, Medsger TA Jr, Hinchcliff M, Hsu V, Wu JY, Fiorentino D, Chung L. Calcinosis is associated with digital ulcers and osteoporosis in patients with systemic sclerosis: A Scleroderma Clinical Trials Consortium study. Semin Arthritis Rheum. 2016 Dec;46(3):344-349. doi: 10.1016/j.semarthrit.2016.05.008. Epub 2016 Jun 2. PMID 27371996
- [Background] Valenzuela A, Baron M, Rodriguez-Reyna TS, Proudman S, Khanna D, Young A, Hinchcliff M, Steen V, Gordon J, Hsu V, Castelino FV, Schoenfeld S, Li S, Wu JY, Fiorentino D, Chung L. Calcinosis is associated with ischemic manifestations and increased disability in patients with systemic sclerosis. Semin Arthritis Rheum. 2020 Oct;50(5):891-896. doi: 10.1016/j.semarthrit.2020.06.007. Epub 2020 Jun 17. PMID 32898758
- [Background] Cruz-Dominguez MP, Garcia-Collinot G, Saavedra MA, Medina G, Carranza-Muleiro RA, Vera-Lastra OL, Jara LJ. Clinical, biochemical, and radiological characterization of the calcinosis in a cohort of Mexican patients with systemic sclerosis. Clin Rheumatol. 2017 Jan;36(1):111-117. doi: 10.1007/s10067-016-3412-9. Epub 2016 Oct 7. PMID 27718018
- [Background] Bartoli F, Fiori G, Braschi F, Amanzi L, Bruni C, Blagojevic J, Bellando-Randone S, Cometi L, de Souza Mueller C, Guiducci S, Rasero L, Epifani F, Furst DE, Matucci-Cerinic M. Calcinosis in systemic sclerosis: subsets, distribution and complications. Rheumatology (Oxford). 2016 Sep;55(9):1610-4. doi: 10.1093/rheumatology/kew193. Epub 2016 May 30. PMID 27241706
- [Background] Gauhar R, Wilkinson J, Harris J, Manning J, Herrick AL. Calcinosis preferentially affects the thumb compared to other fingers in patients with systemic sclerosis. Scand J Rheumatol. 2016 Jul;45(4):317-20. doi: 10.3109/03009742.2015.1127412. Epub 2016 Jan 26. PMID 26812367
- [Background] Valenzuela A, Song P, Chung L. Calcinosis in scleroderma. Curr Opin Rheumatol. 2018 Nov;30(6):554-561. doi: 10.1097/BOR.0000000000000539. PMID 30124603
- [Background] Gorrepati PL, Smith GP. Treatments for calcinosis cutis in autoimmune connective tissue diseases. J Am Acad Dermatol. 2022 Nov;87(5):1211-1212. doi: 10.1016/j.jaad.2022.03.029. Epub 2022 Mar 22. No abstract available. PMID 35331808
- [Background] Nigwekar SU. Multidisciplinary approach to calcific uremic arteriolopathy. Curr Opin Nephrol Hypertens. 2015 Nov;24(6):531-7. doi: 10.1097/MNH.0000000000000175. PMID 26371529
- [Background] Bair B, Fivenson D. A novel treatment for ulcerative calcinosis cutis. J Drugs Dermatol. 2011 Sep;10(9):1042-4. PMID 22052275
- [Background] Goossens J, Courbebaisse M, Caudron E, Bahans C, Vacquerie V, Melchior J, Salle PV, Moesch C, Daudon M, Frocht V, Richette P, Ea HK, Guigonis V. Efficacy of intralesional sodium thiosulfate injections for disabling tumoral calcinosis: Two cases. Semin Arthritis Rheum. 2017 Dec;47(3):451-455. doi: 10.1016/j.semarthrit.2017.05.013. Epub 2017 Jun 17. PMID 28779847
- [Background] Baumgartner-Nielsen J, Olesen AB. Treatment of Skin Calcifications with Intra-lesional Injection of Sodium Thiosulphate: A Case Series. Acta Derm Venereol. 2016 Feb;96(2):257-8. doi: 10.2340/00015555-2206. No abstract available. PMID 26258586
- [Background] Song P, Fett NM, Lin J, Merola JF, Costner M, Vleugels RA. Lack of response to intravenous sodium thiosulfate in three cases of extensive connective tissue disease-associated calcinosis cutis. Br J Dermatol. 2018 Jun;178(6):1412-1415. doi: 10.1111/bjd.15783. Epub 2018 Mar 7. PMID 28667747
- [Background] Mageau A, Guigonis V, Ratzimbasafy V, Bardin T, Richette P, Urena P, Ea HK. Intravenous sodium thiosulfate for treating tumoral calcinosis associated with systemic disorders: Report of four cases. Joint Bone Spine. 2017 May;84(3):341-344. doi: 10.1016/j.jbspin.2016.10.009. Epub 2016 Dec 7. PMID 27955821
- [Background] Del Barrio-Diaz P, Moll-Manzur C, Alvarez-Veliz S, Vera-Kellet C. Topical sodium metabisulfite for the treatment of calcinosis cutis: a promising new therapy. Br J Dermatol. 2016 Sep;175(3):608-11. doi: 10.1111/bjd.14412. Epub 2016 Apr 17. PMID 26799451
- [Background] Patra S, Gupta V, Kumar R, Verma KK. Clinical and radiological improvement in idiopathic calcinosis cutis with topical 25% sodium metabisulfite. Int J Dermatol. 2017 Dec;56(12):1464-1465. doi: 10.1111/ijd.13789. Epub 2017 Oct 26. No abstract available. PMID 29076152
- [Background] Chung L, Valenzuela A, Fiorentino D, Stevens K, Li S, Harris J, Hutchinson C, Assassi S, Beretta L, Lakshminarayanan S, Rodriguez-Reyna TS, Denton CP, Taillefer RG, Herrick AL, Baron M; Scleroderma Clinical Trials Consortium Calcinosis Working Group. Validation of a novel radiographic scoring system for calcinosis affecting the hands of patients with systemic sclerosis. Arthritis Care Res (Hoboken). 2015 Mar;67(3):425-30. doi: 10.1002/acr.22434. PMID 25155948
- [Background] Valenzuela A, Stevens K, Chung MP, Rodriguez-Reyna TS, Proudman S, Baron M, Castelino FV, Hsu V, Green L, Galdo FD, Li S, Fiorentino D, Chung L. Change in calcinosis over 1 year using the scleroderma clinical trials consortium radiologic scoring system for calcinosis of the hands in patients with systemic sclerosis. Semin Arthritis Rheum. 2022 Apr;53:151980. doi: 10.1016/j.semarthrit.2022.151980. Epub 2022 Feb 10. PMID 35183935
- [Background] Gamissans M, Giavedoni P, Roe E, Sanchez J, Quintana-Codina M, Garbayo-Salmons P, Vidal D, Riera-Marti N, Lopez-Llunell C, Romani J, Wortsman X. Multicentric Study on High-Frequency Ultrasound Characterization of Calcium Deposits in Dermal and Subcutaneous Calciphylaxis and Calcinosis. J Ultrasound Med. 2022 Aug;41(8):1975-1979. doi: 10.1002/jum.15878. Epub 2021 Nov 10. PMID 34755910